CLINICAL TRIAL: NCT00475891
Title: Determination of Genetic Relatedness of Linezolid-resistant Vancomycin-resistant Enterococci (VRE) Surveillance Cultures
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: PRO07050007
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Isolate; Linezolid
Keywords: isolate; infection; linezolid
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study will help in identifying the best empiric antibiotic option for Linezolid resistant Vancomycin-resistant Enterococci (VRE) infections. This research is important because it allows the determination of resistance rates to antibiotics that may not be frequently tested to by the clinical microbiology laboratory at UPMC-Presbyterian. It also will provide antibiotic minimum inhibitory concentrations (MICs) for these pathogens which may help in identifying the best empiric antibiotic option for Linezolid-resistant VRE infections.

DETAILED DESCRIPTION:
After 20 linezolid-resistant VRE isolates are identified, genetic relatedness will be determined using a method known as Pulse-field gel electrophoresis (PFGE). No patient related data will accompany these isolates, nor will any related identifiers. These isolates will be tested using standardized susceptibility methods. We will then grow each isolate and test via approved laboratory standards (E-test, AB Biodisk, Stockholm, Sweden) to the drug linezolid. Those determined to be resistant using this approved methodology will be saved until 20 isolates are identified. For resistant isolates found, analytical and molecular techniques will be performed to determine the mechanisms of resistance and whether resistant isolates are coming from a single source/being transmitted from person to person.

ELIGIBILITY:
Inclusion Criteria:

* Dr. Harrison's laboratory collected the rectal surveillance isolates for infection control purposes. The isolates will be from January 1, 2006 to December 31, 2006.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: isolates for rectal surveillance
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-04; Primary Completion 2010-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
dead or alive | end of study
  health status

CONTACTS AND LOCATIONS:
Overall Officials: Brian Potoski, Pharm D, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States